CLINICAL TRIAL: NCT02497131
Title: Phase II Study on the Role of Brentuximab Vedotin as Single Agent in the Treatment of Relapsed/Refractory CD30 Positive Peripheral T Cell Lymphoma (PTCL) Patients
Brief Title: Study on the Role of Brentuximab Vedotin as Single Agent in the Treatment of Relapsed/Refractory CD30+ PTCL Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_PTCL_BV
Record Dates: First submitted 2015-07-08; First posted 2015-07-14 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Lymphatic Diseases
Keywords: PTCL; CD30+
MeSH Terms: conditions — Lymphatic Diseases | interventions — Brentuximab Vedotin

STUDY DESIGN:
Intervention Model Description: Subjects will receive 1.8 mg/kg of brentuximab vedotin as an iv infusion administered on Day 1 of each 21-day cycle for a maximum of 16 cycles.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brentuximab Vedotin 16 cycles (Experimental): Subjects will receive 1.8 mg/kg of brentuximab vedotin as an iv infusion administered on Day 1 of each 21-day cycle for a maximum of 16 cycles.
  Interventions: Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: Brentuximab Vedotin — Brentuximab vedotin will be administered on Day 1 of each 21-day cycle. The dose of brentuximab vedotin is 1.8 mg/kg and is administered by outpatient IV infusion given over approximately 30 minutes
  Other Names: SGN35

SUMMARY:
This is a single-arm, open-label, multicenter, clinical trial to evaluate the efficacy and safety of Brentuximab Vedotin (BV) as a single agent in relapsed/refractory CD30+ PTCL patients.

DETAILED DESCRIPTION:
BV will be administered as a single IV infusion on Day 1 of each 21-day cycle. Measures of anti-cancer activity will be assessed using the revised response criteria for malignant lymphoma (Cheson et al. 2007).

Computed tomography (CT) scans (chest, neck, abdomen, and pelvis) and PET scan will be performed at baseline and Cycles 3, 8, 12, and 16. Patients will have an End of Treatment (EOT) assessment 30 ± 7 days after receiving their final dose of study drug. Patients with at least stable disease will enter short follow up phase till month 24 with radiology assessment every 6 months and visit every 12 weeks. After month 24 and for all patients with progressive disease, long-term follow-up assessments (including survival, disease status and next therapy information) will be performed every 12 weeks until either patient death or study closure, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Males and females ≥18 and ≤75 years at the time of enrolment.
* Histologically confirmed diagnosis of PTCL (PTCL-not otherwise specified [PTCL-NOS], angioimmunoblastic T cell lymphoma [AILT] and transformed mycosis fungoides) according to World Health Organization (2008) classification.
* Histologically confirmed CD30+ PTCL.
* Availability of histological material for central review and pathobiological studies.
* Failed at least one prior systemic antilymphoma therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 1 at study entry.
* At least one site of disease measurable in two dimensions by computed tomography. Both nodal and extranodal disease will be considered (lymphnodes must have long axis of 1.5 cm regardless of short axis or long axis 1.1 to 1.5 cm and short axis >1.0 cm).
* Hematology values within the following limits:

  * Absolute neutrophil count (ANC) ≥ 1500/mm3 independent of growth factor support.
  * Platelets ≥75,000/mm3 or ≥50,000/mm3 if bone marrow involvement is independent of transfusion support.
  * Hemoglobin level ≥8 g/dL.
* Biochemical values within the following limits:

  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3 x upper limit of normal (ULN).
  * Total bilirubin < 1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of nonhepatic origin).
  * Serum creatinine ≤ 2 x ULN.
  * Serum albumin ≥ 3 g/dL.
* Women of childbearing potential (WOCBP) must have a negative pregnancy test within 7 days of receiving study medication.
* WOCBP must agree to use effective contraception, defined as oral contraceptives, double barrier method or practice true abstinence from sexual intercourse during the study and for 6 months after the last dose of study drug.
* Male subjects and their female partners of childbearing potential must be willing to use an appropriate method of contraception or practice true abstinence from sexual intercourse during the study and for 6 months after the last dose of study drug.

Exclusion Criteria:

* Diagnosis of CTCL, ALCL, mycosis fungoides or Sezary Syndrome.
* CD30 expression < 10 %.
* Patients that have not completed any prior treatment chemotherapy and/or other investigational agents within at least 5 half-lives of last dose of that prior treatment.
* Patients underwent major surgery without complete recovery
* Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of brentuximab vedotin.
* Any serious active disease or co-morbid medical condition (according to investigator's decision).
* Prior history of malignancies other than lymphoma (except for a history of a complete resection for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the subject has been free of the disease for ≥ 3 years.
* Patients with peripheral neuropathy of grade 3-4 (also grade 2 with persistent pain, unresponsive to treatment).
* Signs or symptoms of progressive multifocal leukoencephalopathy (PML).
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or lactating females or men or women of childbearing potential not willing to use an adequate method of birth control for the duration of the study.
* CNS disease (meningeal and/or brain involvement by lymphoma) or testicular involvement.
* History of clinically relevant liver or renal insufficiency; significant cardiac, vascular pulmonary, gastrointestinal, endocrine, neurologic, rheumatologic, hematologic, psychiatric, or metabolic disturbances.
* Known history of any of the following cardiovascular conditions:

  * Myocardial infarction within 2 years from enrollment
  * New York Heart Association (NYHA) Class III or IV heart failure
  * Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
  * Recent evidence (within 6 months before first dose of study drug) of a left-ventricular ejection fraction <50%
* Active opportunistic infection.
* Known history of Human Immunodeficiency Virus (HIV) or Hepatitis C or active infection with Hepatitis B.
* Prior allogeneic stem cell transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-09-21 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
overall objective response rate (ORR) | 1 year
  Overall objective response rate (ORR) is defined as the proportion of patients with complete remission (CR) or partial remission (PR) according to the Revised Response Criteria for Malignant Lymphoma

SECONDARY OUTCOMES:
Duration of response | 1 year
  Duration of response is defined as the time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of objective tumor progression or to death due to lymphoma
Complete remission rate (CR) | 1 year
  The proportion of patients with complete remission (CR) according to the Revised Response Criteria for Malignant Lymphoma
Progression-free survival (PSF) | 1 year
  Progression-free survival (PFS) is defined as the time from start of study treatment to first documentation of objective tumor progression or to death due to any cause
Overall survival (OS) | 1 year
  Overall survival (OS) is defined as the time from start of study treatment to date of death due to any cause.
Adverse Events | 1 year
  Type, incidence, severity, seriousness, and relatedness of adverse events, and laboratory abnormalities

OTHER OUTCOMES:
Event-Free survival (EFS) | 1 year
  Event-free survival (EFS) is defined as the time from start of study treatment to any treatment failure including disease progression, or discontinuation of treatment for any reason
B symptom resolution rate | 1 year
  B symptom resolution rate is defined as the proportion of patients with lymphoma-related B symptoms at baseline who achieve resolution of all B symptoms at any time during the treatment period.
CD30 expression | 1 year
  Correlation between CD30 expression and response

CONTACTS AND LOCATIONS:
Overall Officials: Vittorio Stefoni, MD, Principal Investigator — Ematologia "L. & A. Seragnoli" - Policlinico S. Orsola Malpighi
Locations (4):
- Italy (4):
  - Ematologia "L. & A. Seragnoli" - Policlinico S. Orsola Malpighi, Bologna
  - Ematologia e Trapianto IRCCS, Istituto Nazionale dei Tumori, Milan
  - SC Ematologia - Città della Salute e della Scienza, Torino
  - A.O. Universitaria S. Maria Della Misericordia Di Udine, Udine